CLINICAL TRIAL: NCT03372070
Title: Continuous Negative External Pressure (cNEP) for the Treatment of Primary Snoring: A Pilot Study
Brief Title: Continuous Negative External Pressure for the Treatment of Primary Snoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Sommetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOM-026
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Snoring
Keywords: primary snoring; bed partner; home sleep testing
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- cNEP (Experimental): silicone collar applied to anterior neck
  Interventions: Device: cNEP

INTERVENTIONS:
Device: cNEP — soft silicon collar applied to anterior neck with negative pressure
  Other Names: continuous negative external pressure

SUMMARY:
The aim of this pilot study is to gain information on the ability of a continuous negative external pressure collar to safely reduce snoring in primary snorers, and if so to determine whether the reduction in snoring has benefits for both the snorer and the bed partner. This clinical trial will involve both the snorer and his or her bed partner, both of whom must qualify and provide informed consent for participation.

ELIGIBILITY:
Key Snorer Inclusion Criteria:

* BMI <35
* if a previously done polysomnogram (PSG) is available, AHI<5
* snoring identified by a previous PSG and/or by the bed partner

Key bed partner Inclusion criteria

* must have regularly slept with the snorer over the previous month and must plan to sleep with the snorer for the duration of the trial
* considers that the snorer's snoring is a problem
* must discontinue use of any snore-masking equipment or ear plug for at least two weeks prior to the initial visit to the study site and agree to refrain from their use for the duration of the trial

Key snorer exclusion criteria:

* sleep disturbance other than snoring
* snoring due primarily to abnormality of the nasopharynx
* use of snoring treatment during the month prior to the initial visit
* neck anatomic or skin abnormalities
* serious medical condition
* excessive drug or alcohol intake

Key bed partner exclusion criteria:

-known sleep disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
change in snoring duration | two weeks after initiation of treatment
  duration of snoring as a percent of total sleep time compared to baseline

SECONDARY OUTCOMES:
change in apnea-hypopnea index (AHI) | two weeks after initiation of treatment
  mean AHI compared to baseline
change in snoring intensity | two weeks after initiation of treatment
  mean dBC compared to baseline
Treatment-emergent adverse events | two weeks
  tabulation of all adverse events during the clinical trial
change in Epworth Sleepiness Scale (ESS) | two weeks after initiation of treatment
  mean ESS compared to baseline (total range 0-24; lower score means less sleepy)
Short Form Survey 36 (SF-36) | one week time frame, administered two weeks after initiation of treatment
  mean SF-36 compared to baseline
Clinical Global Impression (CGI) Scale: Snorer's sleep | previous week, assessed one and two weeks after initiation of treatment
  CGI "usual sleep score" vs baseline (score range "very much better to very much worse"
Clinical Global Impression (CGI) Scale: Bed partner's complaints about snoring | previous week, assessed one and two weeks after initiation of treatment
  CGI "bed partner complaints about your snoring" scale vs baseline (score range "complained very much less, to "complained very much more"
Clinical Global Impression (CGI) Scale: Acceptability of cNEP | "overall experience to date", assessed one and two weeks after initiation of treatment
  CGI "bed partner complaints about your snoring" scale vs baseline (score range "complained very much less, to "complained very much more"
Clinical Global Impression (CGI) Scale: Bed partner's impression of snorer's sleep | previous week, assessed one and two weeks after initiation of treatment
  CGI scale comparing snorer's sleep to baseline (score range "very much better to very much worse"
Clinical Global Impression (CGI) Scales: bed partner's sleep | previous week, assessed one and two weeks after initiation of treatment
  CGI scale comparing bed partner's sleep to baseline (score range "very much better to very much worse"
Clinical Global Impression (CGI) Scale: Bed partner's overall relationship with snorer | previous week, assessed one and two weeks after initiation of treatment
  CGI scale comparing bed partner's overall relationship wtih snorer to baseline (score range "very much better to very much worse"

CONTACTS AND LOCATIONS:
Overall Officials: Reena Mehra, MD, Principal Investigator — Cleveland Clinic Lerner College of Medicine
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided